CLINICAL TRIAL: NCT04191382
Title: Phase 2 Window Study of Two Dose Levels of Amcenestrant [SAR439859] (SERD) Versus Letrozole in Newly Diagnosed Pre-operative Post-menopausal Patients With ER Positive, HER2 Negative Primary Breast Cancer
Brief Title: Phase 2 Window Study of SAR439859 (Amcenestrant) Versus Letrozole in Post-menopausal Patients With ER+, HER2- Pre-operative Post-menopausal Primary Breast Cancer
Acronym: AMEERA-4
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: early discontinuation based on strategic sponsor decision not driven by any safety concerns
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ACT16106; 2019-002015-26 (EudraCT Number); U1111-1228-9473 (Other: UTN)
Record Dates: First submitted 2019-12-05; First posted 2019-12-09 (Actual); Results first posted 2022-06-29 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Letrozole

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Amcenestrant 400 mg (Experimental): Participants received 4 capsules of 100 milligrams (mg) of amcenestrant once daily (QD) from Day 1 to Day 14.
  Interventions: Drug: Amcenestrant (SAR439859)
- Amcenestrant 200 mg (Experimental): Participants received 2 capsules of 100 mg of amcenestrant QD from Day 1 to Day 14.
  Interventions: Drug: Amcenestrant (SAR439859)
- Letrozole 2.5 mg (Active Comparator): Participants received 2.5 mg of letrozole tablet QD from Day 1 to Day 14.
  Interventions: Drug: Letrozole

INTERVENTIONS:
Drug: Amcenestrant (SAR439859) — Pharmaceutical form: Capsules, Route of administration: Oral
  Arms: Amcenestrant 200 mg; Amcenestrant 400 mg
Drug: Letrozole — Pharmaceutical form: Tablets, Route of administration: Oral
  Arms: Letrozole 2.5 mg

SUMMARY:
Primary Objective:

To determine whether amcenestrant given at 2 different doses improved the antiproliferative activity when compared to letrozole.

Secondary Objectives:

* To assess the proportion of participants with a relative decrease from Baseline in percentage of positive tumor cells tested by immunohistochemistry greater than or equal to (>=) 50 percent (%) (Ki67 >=50%) in the three treatment arms.
* To assess estrogen receptor (ER) degradation in biopsies in participants in the three treatment arms.
* To assess safety in the three treatment arms.

DETAILED DESCRIPTION:
Duration of the study, per participant, would include screening period of up to 14 days before randomization, treatment period of 14 days and post-treatment safety follow-up period of 30±7 days after last investigational medicinal product (IMP) intake.

ELIGIBILITY:
Inclusion criteria :

* Histological or cytological proven diagnosis of invasive breast adenocarcinoma.
* Localized breast cancer eligible for upfront breast conservative surgery or upfront mastectomy: Stage I, Stage II or operable Stage III (excluded T4) as defined in American Joint Committee on Cancer (AJCC) Cancer Staging Manual 8th edition 2017.
* Postmenopausal women as defined by one of the following:
* Spontaneous cessation of menses greater than (>) 12 months.
* or who had received hormonal replacement therapy but had discontinued the treatment and had follicle stimulating hormone (FSH) level in the postmenopausal range.
* or with status post bilateral surgical oophorectomy.
* or post bilateral ovarian ablation through pelvic radiotherapy.
* Breast tumor size of at least 10 millimeters (mm) in greatest dimension measured by ultrasound.
* Primary tumor had to be positive for Estrogen Receptors (ER+) and negative for HER2 (HER2-) receptor by immunohistochemistry.
* Ki67 level of at least 15% at diagnosis from immunohistochemistry of the tumor.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1.

Exclusion criteria:

* Medical history or ongoing gastrointestinal disorders potentially affecting the absorption of SAR439859 or letrozole.
* Participants unable to swallow normally and to take capsules or tablets.
* Participants with known active hepatitis A, B, C infection; or hepatic cirrhosis.
* Participant with any other cancer; adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer or any other cancer from which the participant had been disease free for >3 years were allowed.
* Evidence of metastatic spread by standard assessment according to local practice.
* Treatment with strong Cytochrome P450 3A (CYP3A) inducers or drugs that had the potential to inhibit uridine diphosphate glucuronosyltransferase (UGT) within 2 weeks before first study treatment administration or 5 elimination half-lives whichever was longest.
* Treatment with drugs that were sensitive substrates of P-glycoprotein (P-gp) or of breast cancer resistance protein (BCRP) within 2 weeks before first study treatment administration or 5 elimination half-lives whichever was longer.
* Use of any investigational agent within 4 weeks prior to randomization.
* Recent use of hormone replacement therapy (last dose less than or equal to [<=] 30 days prior to randomization).
* Prior anti-cancer treatment was not allowed unless it was then completed at least 1 year prior to inclusion into this trial.
* Previous systemic or local treatment for the new primary breast cancer currently under investigation (including surgery, radiotherapy, cytotoxic and endocrine treatments).
* Inadequate hematological or renal function.
* Prothrombin time/international normalized ratio (INR) >1.5 * upper limit of normal (ULN) or outside therapeutic range if received anticoagulation that would have had affected the prothrombin time/INR.
* Any of the following abnormal liver function test results: Aspartate aminotransferase >1.5 * ULN; Alanine aminotransferase >1.5 * ULN; Total bilirubin >1.5 * ULN.
* Participants were employees of the clinical study site or other individuals directly involved in the conduct of the study, or immediate family members of such individuals.
* Sensitivity to any of the study interventions, or components thereof, or drug or other allergy that, in the opinion of the Investigator, contraindicates participation in the study.

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2020-02-04 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-05-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (32):
- United States (6):
  - Investigational Site Number 8400014, Tucson, Arizona
  - Investigational Site Number 8400010, Los Angeles, California
  - Investigational Site Number 8400018, Fort Wayne, Indiana
  - Investigational Site Number 8400005, Lincoln, Nebraska
  - Investigational Site Number 8400016, Winston-Salem, North Carolina
  - Investigational Site Number 8400012, Tacoma, Washington
- Belgium (2):
  - Investigational Site Number 0560001, Leuven
  - Investigational Site Number 0560002, Namur
- France (4):
  - Investigational Site Number 2500001, Nantes
  - Investigational Site Number 2500004, Paris
  - Investigational Site Number 2500002, Saint-Cloud
  - Investigational Site Number 2500003, Toulouse
- Italy (3):
  - Investigational Site Number 3800004, Meldola
  - Investigational Site Number 3800002, Milan
  - Investigational Site Number 3800001, Milan
- Japan (3):
  - Investigational Site Number 3920002, Osaka
  - Investigational Site Number 3920003, Sapporo
  - Investigational Site Number 3920001, Yokohama
- Investigational Site Number 8400007, Hato Rey, Puerto Rico
- Russia (5):
  - Investigational Site Number 6430006, Moscow
  - Investigational Site Number 6430004, Moscow
  - Investigational Site Number 6430003, Saint Petersburg
  - Investigational Site Number 6430007, Saint Petersburg
  - Investigational Site Number 6430002, Saint Petersburg
- Spain (4):
  - Investigational Site Number 7240005, Barcelona
  - Investigational Site Number 7240003, Córdoba
  - Investigational Site Number 7240001, Madrid
  - Investigational Site Number 7240002, Valencia
- Ukraine (4):
  - Investigational Site Number 8040004, Kharkiv
  - Investigational Site Number 8040001, Uzhhorod
  - Investigational Site Number 8040002, Vinnytsia
  - Investigational Site Number 8040005, Zaporizhzhya

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Campone M, Bidard FC, Neven P, Wang L, Ling B, Dong Y, Paux G, Herold C, De Giorgi U. AMEERA-4: a randomized, preoperative window-of-opportunity study of amcenestrant versus letrozole in early breast cancer. Breast Cancer Res. 2023 Nov 10;25(1):141. doi: 10.1186/s13058-023-01740-2. PMID 37950338
- See also: ACT16106 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25188&tenant=MT_SNY_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 32 active sites in 8 countries. A total of 135 participants were screened from 04-February-2020 to 21-April-2021, of which 30 participants were screen failures mainly due to selection criteria not met.
Pre-assignment Details: A total of 105 participants with early breast cancer were randomized in 1:1:1 ratio to receive treatment with amcenestrant 400 milligrams (mg), amcenestrant 200 mg, or letrozole 2.5 mg.
Groups:
- Amcenestrant 400 mg: Participants received 4 capsules of 100 mg of amcenestrant once daily (QD) from Day 1 to Day 14.
Period: Overall Study
Arm/Group | Amcenestrant 400 mg | Amcenestrant 200 mg | Letrozole 2.5 mg
Started (Randomized) | 34 | 36 | 35
Treated | 33 | 36 | 35
Completed | 33 | 36 | 35
Not Completed | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Analysis was performed on intent-to-treat (ITT) population that included all enrolled participants for whom there was a confirmation of successful allocation of a randomization number by interactive response technology (IRT) and were analyzed according to the treatment arm assigned at randomization.
Arm/Group | Amcenestrant 400 mg | Amcenestrant 200 mg | Letrozole 2.5 mg | Total Title
Number analyzed (Participants) | 34 | 36 | 35 | 105
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.4 (8.6) | 63.4 (8.4) | 63.7 (8.5) | 63.2 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 36 | 35 | 105
  Male | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 3 | 5 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1
  White | 23 | 24 | 25 | 72
  More than one race | 0 | 1 | 1 | 2
  Unknown or Not Reported | 8 | 8 | 4 | 20
Ki67 expression at Baseline [Mean (Standard Deviation); unit: percentage of positive tumor cells] — Tumor tissue collected through a core-cut biopsy at Baseline was used to determine Ki67 expression. Ki67 expression was defined as the percentage of positive tumor cells assessed by central reading. Population: Here, 'Number analyzed' signifies participants with available data at Baseline for the specified Baseline measure.
  percentage of positive tumor cells
    number analyzed (Participants) | 32 | 36 | 32 | 100
    (all) | 33.8 (16.3) | 31.2 (14.3) | 32.6 (18.5) | 32.5 (16.3)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Ki67 Level at Day 15
Description: Tumor tissue collected through a core-cut biopsy at Baseline and Day 15 was used to determine Ki67 expression. Ki67 expression was defined as the percentage of positive tumor cells assessed by central reading. Ki67 percent change from Baseline for a given participant was defined as 100*(Ki67pre - Ki67post) / Ki67pre, where Ki67pre and Ki67post were pre-treatment and post-treatment Ki67 value of the participant. Adjusted geometric least square (LS) means and 95 percentage (%) confidence interval (CI) for the percent change were obtained from analysis of covariance (ANCOVA) model of the log proportional change i.e., log (Ki67post/ki67pre) with treatment and log-Ki67pre as fixed effect and converted by antilog transformation.
Time Frame: Baseline, Day 15
Population: Analysis was performed on modified intent-to-treat (mITT) population that included all enrolled participants for whom there was a confirmation of successful allocation of a randomization number by IRT, who had taken at least one study drug, and who had both Baseline and post treatment available biopsies with Ki67 values.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Amcenestrant 400 mg | Amcenestrant 200 mg | Letrozole 2.5 mg
Number analyzed (Participants) | 31 | 35 | 29
percent change | 75.9 [67.9 to 81.9] | 68.2 [58.4 to 75.7] | 77.7 [70.0 to 83.4]
Statistical Analysis 1: Comparison: Amcenestrant 400 mg vs Letrozole 2.5 mg; Geometric LS-means ratio of proportional change was the ratio of geometric LS-means of the proportional change between groups (Amcenestrant 400 mg versus Letrozole 2.5 mg); Test type: Other — Other descriptive analysis; Ratio of Geometric Means = 1.08, 95% CI 2-sided [0.72 to 1.63]
Statistical Analysis 2: Comparison: Amcenestrant 200 mg vs Letrozole 2.5 mg; Geometric LS-means ratio of proportional change was the ratio of geometric LS-means of the proportional change between groups (Amcenestrant 200 mg versus Letrozole 2.5 mg); Test type: Other — Other descriptive analysis; Ratio of Geometric Means = 1.42, 95% CI 2-sided [0.95 to 2.12]

2. Secondary Outcome: Percentage of Participants With Percent Change From Baseline in Ki67 Greater Than or Equal to (>=) 50 Percent at Day 15
Description: Tumor tissue collected through a core-cut biopsy at Baseline and Day 15 was used to determine Ki67 expression. Ki67 expression was defined as the percentage of positive tumor cells assessed by central reading. Ki67 percent change from Baseline for a given participant was defined as 100*(Ki67pre - Ki67post) / Ki67pre, where Ki67pre and Ki67post were pre-treatment and post-treatment Ki67 value of the participant.
Time Frame: Baseline, Day 15
Population: Analysis was performed on mITT population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Amcenestrant 400 mg | Amcenestrant 200 mg | Letrozole 2.5 mg
Number analyzed (Participants) | 31 | 35 | 29
percentage of participants | 74.2 [55.4 to 88.1] | 68.6 [50.7 to 83.1] | 89.7 [72.6 to 97.8]

3. Secondary Outcome: Change From Baseline in Estrogen Receptor (ER) Expression as Measured by H-Score at Day 15
Description: Change from Baseline in ER expression was measured by H-Score. The H-score was calculated as the sum of the percent of cells staining positive (0 to 100) multiplied staining intensity level from 0 to 3 (0=none, 1=low, 2=moderate, 3=high). Total ER expression H-score ranged from 0 to 300, where higher score indicated stronger ER expression. Change from Baseline in H-Score equals H-scorepost minus H-scorepre; where H-scorepost and H-scorepre denoted post-treatment and pre-treatment H-scores, respectively. LS-means and 95% CI were obtained from an ANCOVA model for change from baseline with treatment and baseline as fixed effect.
Time Frame: Baseline, Day 15
Population: Analysis was performed on mITT population. Here, 'overall number of participants analyzed' signifies participants with available data for this outcome measure.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Amcenestrant 400 mg | Amcenestrant 200 mg | Letrozole 2.5 mg
Number analyzed (Participants) | 28 | 32 | 28
score on a scale | -176.7 [-201.4 to -152.0] | -202.9 [-226.1 to -179.7] | -32.5 [-57.2 to -7.7]

4. Secondary Outcome: Number of Participants With Abnormalities: Hematological Parameters
Description: Hematology parameters covered by National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) and included: Hemoglobin, Lymphocyte, Neutrophils, Leukocytes (white blood cells), Anemia, Platelets, Eosinophils, and international normalized ratio (INR). An NCI-CTCAE Grades 1 to 5 were described as: Grade 1-Mild; asymptomatic/mild symptoms; Grade 2-Moderate; minimal, local or noninvasive intervention indicated; limiting age appropriate instrumental daily activities. Grade 3-Severe/medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; Grade 4-Life-threatening consequences; Grade 5-Death. Data for 'All Grades' were reported in this outcome measure.
Time Frame: From first dose of study drug up to Day 14
Population: Analysis was performed on safety population that included all participants who were randomly assigned to study drug and who took at least 1 dose of study drug. Here, 'Number analyzed' signifies participants with available data for each specified category for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Amcenestrant 400 mg | Amcenestrant 200 mg | Letrozole 2.5 mg
Number analyzed (Participants) | 33 | 36 | 35
Participants
  White blood cell decreased: number analyzed (Participants) | 32 | 35 | 35
  White blood cell decreased | 5 | 6 | 3
  Neutrophil count decreased: number analyzed (Participants) | 32 | 35 | 35
  Neutrophil count decreased | 1 | 0 | 1
  Anemia (hemoglobin decreased): number analyzed (Participants) | 32 | 35 | 35
  Anemia (hemoglobin decreased) | 6 | 4 | 1
  Hemoglobin increased: number analyzed (Participants) | 32 | 35 | 35
  Hemoglobin increased | 0 | 0 | 0
  Platelet count decreased: number analyzed (Participants) | 32 | 35 | 35
  Platelet count decreased | 1 | 1 | 0
  Lymphocyte count decreased: number analyzed (Participants) | 32 | 35 | 35
  Lymphocyte count decreased | 1 | 3 | 1
  INR increased: number analyzed (Participants) | 28 | 28 | 31
  INR increased | 0 | 0 | 0
  Eosinophilia (eosinophils increased): number analyzed (Participants) | 32 | 35 | 35
  Eosinophilia (eosinophils increased) | 2 | 1 | 1

5. Secondary Outcome: Number of Participants With Abnormalities: Clinical Chemistry
Description: Clinical chemistry laboratory parameters covered by NCI-CTCAE and included: Glucose, Potassium, Sodium, Creatinine. An NCI-CTCAE Grades 1 to 5 were described as: Grade 1-Mild; asymptomatic or mild symptoms; Grade 2- Moderate; minimal, local or noninvasive intervention indicated; limiting age appropriate instrumental daily activities; Grade 3-Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; Grade 4-Life-threatening consequences; Grade 5-Death. Data for 'All Grades' were reported in this outcome measure.
Time Frame: From first dose of study drug up to Day 14
Population: Analysis was performed on safety population. Here, 'Number analyzed' signifies participants with available data for each specified category for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Amcenestrant 400 mg | Amcenestrant 200 mg | Letrozole 2.5 mg
Number analyzed (Participants) | 33 | 36 | 35
Participants
  Hypernatremia (sodium increased): number analyzed (Participants) | 32 | 35 | 35
  Hypernatremia (sodium increased) | 1 | 1 | 1
  Hyponatremia (sodium decreased): number analyzed (Participants) | 32 | 35 | 35
  Hyponatremia (sodium decreased) | 0 | 1 | 0
  Hyperkalemia (potassium increased): number analyzed (Participants) | 32 | 35 | 35
  Hyperkalemia (potassium increased) | 2 | 1 | 1
  Hypokalemia (potassium decreased): number analyzed (Participants) | 32 | 35 | 35
  Hypokalemia (potassium decreased) | 0 | 2 | 0
  Creatinine increased: number analyzed (Participants) | 32 | 34 | 35
  Creatinine increased | 0 | 3 | 2
  Hypoglycemia (glucose decreased): number analyzed (Participants) | 32 | 35 | 35
  Hypoglycemia (glucose decreased) | 0 | 1 | 0

ADVERSE EVENTS:
Time Frame: From first dose up to 30 days following the last dose of study drug (up to 45 days)
Description: Reported adverse events (AEs) are treatment-emergent adverse events (TEAEs) i.e., AEs that developed, worsened, or became serious during the treatment period (time from the first dose of study drug up to 30 days after last dose of study drug). Analysis was performed on safety population.
Arm/Group | Amcenestrant 400 mg | Amcenestrant 200 mg | Letrozole 2.5 mg
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/36 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/33 | 2/36 | 0/35
Other Adverse Events (participants affected / at risk) | 11/33 | 12/36 | 14/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Amcenestrant 400 mg (N=33) | Amcenestrant 200 mg (N=36) | Letrozole 2.5 mg (N=35)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Wound Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Amcenestrant 400 mg (N=33) | Amcenestrant 200 mg (N=36) | Letrozole 2.5 mg (N=35)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 3 (3) | 3 (3)
Asthenia (General disorders) | 2 (2) | 2 (2) | 0 (0)
Fatigue (General disorders) | 2 (2) | 1 (1) | 1 (1)
Feeling Cold (General disorders) | 2 (2) | 0 (0) | 0 (0)
Procedural Pain (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 2 (2)
Alanine Aminotransferase Increased (Investigations) | 1 (1) | 2 (2) | 0 (0)
Decreased Appetite (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 3 (3)
Headache (Nervous system disorders) | 3 (3) | 0 (0) | 2 (2)
Anxiety (Psychiatric disorders) | 1 (1) | 2 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 4 (4) | 1 (1) | 0 (0)
Breast Pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 3 (3)
Hot Flush (Vascular disorders) | 4 (4) | 1 (1) | 5 (5)

LIMITATIONS AND CAVEATS:
The study recruitment discontinued early based on strategic sponsor decision that was not driven by any safety concerns. No inferential statistical analysis was performed due to early termination.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2021-02-04): https://cdn.clinicaltrials.gov/large-docs/82/NCT04191382/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-09): https://cdn.clinicaltrials.gov/large-docs/82/NCT04191382/SAP_001.pdf